CLINICAL TRIAL: NCT00083304
Title: A Phase 3 Randomized, Open-label Comparative Study of Standard Whole Brain Radiation Therapy With Supplemental Oxygen, With or Without Concurrent RSR13 (Efaproxiral), in Women With Brain Metastases From Breast Cancer
Brief Title: Whole Brain Radiation Therapy With Oxygen, With or Without RSR13, in Women With Brain Metastases From Breast Cancer
Acronym: ENRICH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Medical Monitor, Allos Therapeutics, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-016
Record Dates: First submitted 2004-05-18; First posted 2004-05-19 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Metastases
Keywords: Breast; Brain; RSR13; efaproxiral; Whole Brain Radiation Therapy; Brain metastases; Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — efaproxiral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efaproxiral + WBRT + Supplemental Oxygen (Experimental)
  Interventions: Drug: Efaproxiral; Radiation: Whole Brain Radiation Therapy (WBRT); Other: Supplemental Oxygen
- WBRT + Supplemental Oxygen (Active Comparator)
  Interventions: Radiation: Whole Brain Radiation Therapy (WBRT); Other: Supplemental Oxygen

INTERVENTIONS:
Drug: Efaproxiral — 75 mg/kg, administered over 30 minutes via a central venous access device (CVAD).
  Administered 30 minutes prior to the start of whole brain radiation therapy (WBRT) on each WBRT treatment day for 10 days.
  Other Names: RSR13
  Arms: Efaproxiral + WBRT + Supplemental Oxygen
Radiation: Whole Brain Radiation Therapy (WBRT) — 3.0 Gy per day for 10 days (30.0 Gy total) of WBRT.
Other: Supplemental Oxygen — 4 L/minute by nasal cannula.
  Administered at least 35 minutes prior to WBRT, during WBRT and until 15 minutes after completion of WBRT on all WBRT treatment days.

SUMMARY:
RSR13 (efaproxiral) is a radiation sensitizer that has shown positive results in a Phase 3, randomized clinical trial of patients with brain metastases. Of 111 eligible breast cancer patients with brain metastases in that trial, 59 patients who received RSR13 prior to radiation therapy had a median survival time that was twice as long as the 52 patients who did not receive RSR13 prior to radiation therapy.

RSR13 (efaproxiral) is an experimental drug that increases the amount of oxygen released from blood into the tissues. It is well known that certain types of cancer tumors, including those in brain metastases, lack oxygen. Lack of oxygen in a tumor can reduce the effect of radiation therapy (RT). RSR13 may increase the oxygen level in brain tumors so that radiation therapy works better.

This study will enroll up to 360 women with brain metastases from breast cancer, and will evaluate if whole brain radiation therapy given with RSR13 will have a better treatment effect than whole brain radiation therapy alone. RSR13 will be infused intravenously (IV) through a central catheter placed in a central vein. Women randomized (assigned) to receive RSR13, therefore, will need to have a central catheter placed for treatment unless one is already in place.

DETAILED DESCRIPTION:
The screening process will include documentation of the cancer, which which will require a brain scan and may include a liver scan. Other screening measurements will include a Karnofsky Performance Status (KPS) assessment, measurement of the amount of oxygen in the blood, using a non-invasive device most often placed on the finger, lung function tests that will require blowing into a machine, and an electrocardiogram (ECG). About 2 teaspoons, or 10 mL, of blood will be taken for specific laboratory tests, and a pregnancy test will be done on the blood of women of childbearing potential.

All study patients will receive supplemental oxygen and whole brain radiation therapy (WBRT) (30 Gy, 3 Gy fractions) every weekday for 2 weeks. Half of the patients will be randomized (assigned) to receive RSR13 prior to WBRT, and will need to have a central catheter placed for treatment unless one is already in place. Patients who receive RSR13 will also need to continue to receive oxygen in the clinic until the amount of oxygen in their blood is near normal. This level has returned to near normal in most patients within 1 to 2 hours.

During treatment and follow-up visits, physical and neurological exam, KPS assessment, weight, height, and vital sign measurements, and about 2 teaspoons of blood may be required. Patients will need to return for follow-up visits 1 month after completion of treatment, 2 months later, and every 3 months thereafter until their doctor tells them otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with brain metastases from breast cancer
* Minimum KPS of 70

Exclusion Criteria:

* Previous treatment for brain metastases, including brain surgery and any form of radiation to the brain

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2004-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Measured from randomization until death due to any cause.

SECONDARY OUTCOMES:
Response Rate in the Brain at 3 Months | Assessed at screening, 3 months after end of study treatment and at least 4 weeks after the 3-month scan.
Karnofsky Performance Status & Neurological Signs & Symptoms | Assessed at baseline, 1 month follow-up (FU) visit, 3 month FU visit, and 6 month FU visit.

CONTACTS AND LOCATIONS:
Overall Officials: John Suh, MD, Study Chair — The Cleveland Clinic
Locations (94):
- United States (39):
  - Virginia G. Piper Cancer Center, Arizona Oncology Services, Phoenix, Arizona
  - Arizona Cancer Center, University of Arizona, Tucson, Arizona
  - The University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - University of California at Los Angeles, Los Angeles, California
  - Radiological Associates of Sacramento, Sacramento, California
  - UCSF - Comprehensive Cancer Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Boca Raton Community Hospital, Boca Raton, Florida
  - University of Miami Medical, Miami, Florida
  - University of South Florida - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Maryland Hematology Oncology, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - University of North Carolina Breast Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Division of Hematology-Oncology, Cincinnati, Ohio
  - Cleveland Clinic Hospital, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - Virginia Mason Cancer Center, Seattle, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (5):
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires, Cuidad de Buenos Aires
  - Instituto de Oncologia A. Roffo, Buenos Aires
  - Hospital Espanol, Buenos Aires
  - Instituto Privado de Radioterapia y Oncologia, Córdoba
  - Centro de Terapia Radiante Cumbres (CAICI), Rosario
- Austria (2):
  - LKH-Universitatsklinikum Graz, Graz
  - Medical University Innsbruck, Innsbruck
- Brazil (6):
  - Hospital Sao Lucas PUC, Teófilo, Fortaleza Ceara
  - Fundação Pio XII - Hospital do Câncer de Barretos, Barretos, São Paulo
  - Hospital Erasto Gaertner, Curitiba
  - Velindre Hospital, Porto Alegre
  - Hospital Santa Rita da Irmandade da Santa Casa, Porto Alegre
  - Instituto Brasileiro de Controle do Cancer, São Paulo
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Center, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Campus Notre Dame, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Hotel-Dieu de Quebec du CHUQ, Québec, Quebec
  - Centre Hospitalier Universitarie de Service de Radio-Oncologie, Sherbrooke, Quebec
- Cilnica Santa Maria, Providencia, Santiago de Chile, Chile
- Croatia (3):
  - Clinical Hospital Osijek, Osijek
  - CHU Zagreb University School of Medicine, Zagreb
  - University Hospital for Tumors, Zagreb
- France (10):
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hopital de Montbeliard, Montbéliard
  - Centre Antioned Lacasagne, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Clinique Armoricaine de, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Institut Gustave Roussy, Villejuif
- Hygeia Diagnostic and Therapeutic Center of Athens, Athens, Greece
- Hungary (2):
  - University of Debrecen, Debrecen, Hajdú-Bihar
  - University of Szeged, Szeged
- Italy (2):
  - Azienda Ospedaliera Maggiore della Carita, Novara
  - Ospedale S Chiara, University of Pisa, Pisa
- Lithuania (2):
  - Kaunas Medical University Hospital, Kaunas
  - Institute of Oncology, Vilnius University, Vilnius
- Peru (3):
  - Hospital Edgardo Rebagliati Martins (ESSALUD), Lima
  - Radiooncologia, Radiation Oncology Center, Lima
  - Instituto de Enfermedades Neoplasicas (INEN), Lima
- Spain (5):
  - Instituto Catalan de Oncologia (ICO), Barcelona
  - Ciutat Sanitari de Vall d'Hebron, Barcelona
  - Hospital Ramon Y Cajal, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Instituto Valenciano de Oncologia, Valencia
- United Kingdom (3):
  - Velindre Hospital, Whitchurch, Cardiff
  - Royal Sussex County Hospital, Brighton
  - Beatson Oncolgy Center, Glasgow